CLINICAL TRIAL: NCT05263830
Title: Evaluation of the Contribution of Glypican-3 as a Pronostic Factor in Patients With Advanced Hepatocellular Carcinoma Treated by Immunotherapy
Brief Title: Glypican-3 as a Prognostic Factor in Patients With Hepatocellular Carcinoma Treated by Immunotherapy
Acronym: IMMUNOGLYPIC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210978
Record Dates: First submitted 2022-01-27; First posted 2022-03-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Glypican 3; Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Simpson-Golabi-Behmel syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with hepatocellular carcinoma treated with Atezolizumab / Bevacizumab: Patients with an indication for treatment with Atezolizumab / Bevacizumab for the management of an advanced disciplinary hepatocellular carcinoma in a multidisciplinary consultation meeting.
  Interventions: Other: Quantitative assay of GlypicanPC-3
- Patient with hepatocellular carcinoma treated with Durvalumab/Trémélimumab: Patients with an indication for treatment with Durvalumab/Trémélimumab for the management of an advanced disciplinary hepatocellular carcinoma in a multidisciplinary consultation meeting.
  Interventions: Other: Quantitative assay of GlypicanPC-3

INTERVENTIONS:
Other: Quantitative assay of GlypicanPC-3 — Quantitative assay of GlypicanPC-3 in human serum is performed by direct sandwich immunoassay ( CanAg Glypican3 EIA - Fujirebio ) on microplate using two mouse monoclonal antibodies against two epitopes of the Glypican-3 core protein

SUMMARY:
Recently, the positive results of the Imbrave 150 study (randomized study comparing Atezolizumab+Bevacizumab versus Sorafenib) prompted investigators to redefine their management strategy for advanced HCC by proposing the combination Atezolizumab+ Bevacizumab as first-line treatment in these patients. Identifying new predictive biomarkers of response is essential to optimize the identification of patients who will benefit from immunotherapy. Glypican-3 (GPC-3) is a cell surface glycoprotein that belongs to the family of heparan sulfate chain proteoglycan that is directly implicated in several cancers and more particularly in HCC. GPC-3 overexpression in serum predicts a poor prognosis for patients with HCC and is associated with early tumor recurrence. Through this study, the investigators want to determine whether the concentration of circulating GPC-3 alone, or in combination with other biomarkers used in current practice (PIVKA, AFP) could predict the response to treatment with Atezolizumab/Bevacizumab and OS.

DETAILED DESCRIPTION:
When hepatocellular carcinoma (HCC) is diagnosed, only 25% of patients will be able to have a curative treatment such as liver transplantation, treatment by ablation or surgical resection. In the majority of cases, patients will only have access to so-called palliative treatment. For many years, the only treatment available for patients with advanced HCC was sorafenib, a tyrosine kinase inhibitor with an average overall survival of 10.6 months. Recently, the positive results of the Imbrave 150 study (randomized study comparing Atezolizumab + Bevacizumab versus Sorafenib) prompted investigators to redefine their management strategy for advanced HCC by proposing the combination Atezolizumab+Bevacizumab as first-line treatment in these patients. Indeed, the overall survival (OS) and progression-free survival rates (PFS) were significantly higher in the Atezolizumab+Bevacizumab arm (OS: 67.2% at 12 months and PFS: 6.8 months) versus Sorafenib (OS: 54.6% at 12 months, PFS 4.3 months). The recent approval of the treatment in France is a unique opportunity to carry out a pilot study on clinical, biological, histological, molecular and immune prognostic and predictive factors in patients treated with the Atezolizumab+Bevacizumab combination. Identifying new predictive biomarkers of response is essential to optimize the identification of patients who will benefit from immunotherapy. HCCs are characterized by multiple genomic alterations and the abnormal expression of numerous pro- and anti-oncogenic genes. Glypican-3 (GPC-3) is a cell surface glycoprotein that belongs to the family of heparan sulfate chain proteoglycans. As a co-receptor, GPC-3 is involved in the control of several major signaling pathways (IGF2, Wnt/beta-catenin, etc.) and plays an important role in cell proliferation and tissue growth. At the tumoral level, GPC-3 is directly implicated in several cancers and more particularly in HCC. GPC-3 is overexpressed in 72% of HCCs and its expression is absent in normal liver tissues and benign liver lesions. GPC-3 overexpression is associated with the state of cell tumor differentiation and proliferation in HCC, tumor aggressiveness, as well as poor prognosis and shorter OS. GPC-3 overexpression in serum also predicts a poor prognosis for patients with HCC and is associated with early tumor recurrence. Through this study, the investigators want to determine whether the concentration of circulating GPC-3 alone, or in combination with other biomarkers used in current practice (PIVKA, AFP) could predict the response to treatment with Atezolizumab/Bevacizumab and OS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age < 90 years
* Diagnosed with HCC developed on a cirrhotic liver or on chronic liver disease that has not reached the stage of cirrhosis regardless of the etiology diagnosed according to the diagnostic criteria for TNCD updated in June 2021 (1)
* Having an indication for systemic therapy with Atezolizumab+Bevacizumab validated in multidisciplinary meeting according to the current recommendations of cancer societies.
* Understanding the French language.
* Having been informed and accepted to participate to the study.

Exclusion Criteria:

* HIV or known immune deficiency or immunosuppressive treatment
* Autoimmune diseases or other immunotherapies
* History of portosystemic shunt or liver transplantation
* Sepsis, vasoconstrictor drugs.
* Pregnant or breastfeeding women
* Protected populations: under guardianship or curators

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for treatment with Atezolizumab/Bevacizumab for advanced HCC at a multidisciplinary consultation meeting
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2029-09-08 (Estimated); Study Completion 2029-09-08 (Estimated)

PRIMARY OUTCOMES:
evaluate concentration of circulating GPC-3 | at inclusion, at 3 weeks and at 3 months of the first infusion of Atezolizumab/Bevacizumab
  Evaluation of the change in GPC-3 concentration before, at 3 weeks (second infusion) and at 3 months from the first infusion of Atezolizumab/Bevacizumab .

SECONDARY OUTCOMES:
Evaluate overall survival | at 24 months
Evaluation of the combination of circulating GPC-3 level with other biomarkers (PIVKA, AFP) before, 3 weeks and 3 months after initiation of Atezolizumab/Bevacizumab and/or their variation value could predict treatment response. | at inclusion, at 3 weeks and at 3 months of the first infusion of Atezolizumab/Bevacizumab
  Correlation of the values of GPC-3, PIVKA, AFP
Evaluation of the combination of circulating GPC-3 level with other biomarkers (PIVKA, AFP) before, 3 weeks and 3 months after initiation of Atezolizumab/Bevacizumab and/or their variation value could predict overall Survival. | at inclusion, at 3 weeks and at 3 months of the first infusion of Atezolizumab/Bevacizumab, at 24 months
  Correlation between survival at 24 months and the values of GPC-3, PIVKA, AFP before, 3 weeks and 3 months after the start of treatment and the change in value.
Evaluation of the HCC response to treatment on Imaging assessment (CT-scan and MRI) every 3 months according to the miRECIST criteria (combination of mRECIST and iRECIST criteria) | at inclusion, at 3,6,9,12,15,18,21 and 24 months of the first infusion of Atezolizumab/Bevacizumab,

CONTACTS AND LOCATIONS:
Overall Officials: Manon ALLAIRE, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service hépato-gastroentérologie, Hôpital la Pitié-Salpêtrière, Paris, France